CLINICAL TRIAL: NCT04582617
Title: COSMOS Web: Investigating the Effects of Cocoa Flavanol on Cognition Assessed Online
Brief Title: Investigating the Effects of Cocoa Flavanol on Cognition Assessed Online
Acronym: COSMOS-Web
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Brigham and Women's Hospital (Other); Fred Hutchinson Cancer Center (Other); Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: AAAQ8029
Record Dates: First submitted 2019-10-02; First posted 2020-10-09 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Aging; Cognitive Change
Keywords: Cognitive Function; Cognitive Change; Aging; ModRey; Cocoa Extract; Multivitamin; Hippocampus; Executive Function; Verbal Memory; Spatial Memory
MeSH Terms: interventions — Chocolate; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cocoa extract + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Cocoa Extract; Dietary Supplement: Multivitamin
- Cocoa extract + multivitamin placebo (Active Comparator)
  Interventions: Dietary Supplement: Cocoa Extract; Dietary Supplement: Multivitamin placebo
- Cocoa extract placebo + multivitamin (Active Comparator)
  Interventions: Dietary Supplement: Cocoa Extract Placebo; Dietary Supplement: Multivitamin
- Cocoa extract placebo + multivitamin placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Cocoa Extract Placebo; Dietary Supplement: Multivitamin placebo

INTERVENTIONS:
Dietary Supplement: Cocoa Extract — 2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine
  Arms: Cocoa extract + multivitamin; Cocoa extract + multivitamin placebo
Dietary Supplement: Cocoa Extract Placebo — Cocoa extract placebo
  Arms: Cocoa extract placebo + multivitamin; Cocoa extract placebo + multivitamin placebo
Dietary Supplement: Multivitamin — Multivitamin
  Arms: Cocoa extract + multivitamin; Cocoa extract placebo + multivitamin
Dietary Supplement: Multivitamin placebo — Multivitamin placebo
  Arms: Cocoa extract + multivitamin placebo; Cocoa extract placebo + multivitamin placebo

SUMMARY:
The COcoa Supplement and Multivitamin Outcomes Study (COSMOS; NCT02422745) is a randomized clinical trial of cocoa extract supplement (containing a total of 500 mg/d flavanols, including 80 mg (-)-epicatechin), and/or a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among men aged 60 years and older and women aged 65 years and older. This ancillary study (COSMOS Web) is being conducted among a subset of participants in COSMOS and will examine whether the cocoa extract supplements affects cognitive function in older adults.

DETAILED DESCRIPTION:
The goal of the COSMOS Web study is to determine whether a dietary intervention with flavanol-containing cocoa extract has an effect on cognitive function in older adults (age 60+). The study will be conducted in a subset of 4000 participants from the COSMOS study (NCT02422745). The investigators' recent work (Sloan et al., submitted) showed that cocoa flavanol consumption over 12 weeks led to improvements in immediate recall on the ModRey verbal memory task in healthy older adults.

In COSMOS Web, the investigators are testing the effect of a dietary intervention with flavanol-containing cocoa extract on a range of aging-related cognitive measures, as assessed through a novel online-administered test battery, in a cohort of older participants. Change in ModRey (Modified Rey Auditory Verbal Learning Test) immediate recall performance over 1 year of cocoa extract consumption will be our primary outcome measure. Secondary endpoints will include change in ModRey performance at 2- and 3-year follow-up, and change in performance tests of a novel object recognition task, executive function/working memory, and spatial memory at 1-, 2-, and 3- years follow-up. This study will explore whether baseline measures of cognition and nutritional status can predict differential effects of the cocoa extract supplementation. This study will also explore the effect of multivitamin intake on the primary and secondary outcomes noted above and test whether multivitamin intake interacts with flavanol intake from cocoa extract to enhance or mitigate effects on cognitive outcomes. In a subset of participants evaluated in person, this study will examine the impact of cocoa extract intake and explore the main and interacting effects of multivitamins on cognitive changes and brain structure and function appreciated with magnetic resonance imaging over a 2-year period.

Leveraging the COSMOS study, which has randomized 21,442 older adult participants into cocoa extract and placebo interventions, the study team at Brigham and Women's Hospital, who administer the parent COSMOS trial, are recruiting ~4000 older adult volunteers to participate in COSMOS Web (this study) an online cognitive testing battery developed by the team at Columbia University. These 4000 participants will complete an initial online cognitive assessment and additional assessments after one, two, and three years of follow-up. In addition, approximately 200 COSMOS Web participants who live in the Boston area will complete clinic-based study visits at the Clinical and Translational Science Center at Brigham and Women's Hospital. During that visit, they will complete a neuropsychological test battery, for comparison to their performance online. This study will examine the impact of dietary interventions with cocoa extract and explore the main and interacting effects of multivitamin intake on cognitive changes and brain structure and function appreciated with magnetic resonance imaging over a 2-year period.

After the COSMOS trial began, an advanced method to analyze cocoa flavanols was accredited by AOAC International as a First Action Official Method of Analysis (https://doi.org/10.1093/jaoacint/qsaa132). This updated method relies on a reference material (RM8403) recently standardized and made commercially available by the U.S. National Institute of Standards and Technology. While the actual cocoa flavanol content of the COSMOS intervention remained unchanged throughout the trial, the application of this new analytical method led to expected changes in how the total cocoa flavanol content is now reported. Applying AOAC 2020.05/RM8403 to the COSMOS intervention, the total cocoa flavanol content of the COSMOS intervention is now 500 mg/day. Reporting of (-)-epicatechin content remained unaffected. Going forward, we will therefore apply AOAC 2020.05/RM8403 and report that the COSMOS intervention tested 500 mg/day of cocoa flavanols, including 80 mg of (-)-epicatechin.

ELIGIBILITY:
Participants in COSMOS (NCT02422745) who meet the following criteria are eligible to participate in this ancillary study:

Inclusion Criteria:

* Willingness to participate
* Email and internet access via computer

Exclusion Criteria:

* Analog to COSMOS parent trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3959 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ModRey: 1-Year Change in Immediate Recall/Learning/Episodic Memory | 1-year follow-up
  A measure of verbal memory. The change in the number of words recalled immediately on the ModRey task (Hale et al., 2019), after one year of cocoa extract/placebo intervention.

SECONDARY OUTCOMES:
ModRey: Longitudinal Change in Immediate Recall/Learning | 2-year and 3-year follow-ups
  A measure of verbal memory. Change in number of words recalled immediately on the ModRey task.
ModBent | 1-year, 2-year and 3-year follow-ups
  A measure of pattern separation/object recognition. Change in the mean response time on correct rejection trials on a delayed recognition task.
Flanker: Directional Flanker Effect | 1-year, 2-year and 3-year follow-ups
  A measure of executive control. Change in the difference in reaction time (in ms) between directionally congruent and directional incongruent trials in a Flanker task.
Spatial Reconstruction: Distortion | 1-year, 2-year and 3-year follow-ups
  A measure of spatial memory. Change in the proportion of stimulus pairs where their relative locations are reconstructed differently than originally shown
Self-Reported Memory Change | 1-year, 2-year and 3-year follow-ups
  Self-report of memory change in the last year, on a scale of 1-7
In-clinic ModBent | 2-year follow-up
  Change in performance on the ModBent task, administered in-clinic to a subset of 200 participants
Interaction of Baseline Diet & Intervention on the ModRey | 1-year, 2-year and 3-year follow-ups
  Interaction of baseline diet (as assessed by the Food Frequency Questionnaire) with the flavanol/multivitamin interventions on the ModRey, a measure of verbal memory (change in number of words recalled)
Hippocampal volume change | 2-year follow-up
  Change in hippocampus volume (in cubic mm) in subset of participants with in-clinic MRI scan
Global cortical thickness change | 2-year follow-up
  Change in average cortical thickness in the whole brain (in mm) in subset of participants with in-clinic MRI scan
Hippocampal cerebral blood volume change | 2-year follow-up
  Change in cerebral blood volume in the hippocampus (in cubic mm) in subset of participants with in-clinic MRI scan
Proportions of words recalled on in-clinic list learning task | 2-year follow-up
  Proportions of words recalled on list learning task for subset of participants with in-clinic cognitive testing

CONTACTS AND LOCATIONS:
Overall Officials: Adam M. Brickman, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in study data may contact the study principal investigators to request access. Data requests must be submitted in writing for approval by qualified individuals; they will be reviewed by study investigators. External investigators who are granted access to data for analysis must identify a Cosmos Web investigator, who will participate in analyses and manuscript preparation as a co-author. Researchers interested in accessing data related to the Cosmos parent trial (NCT02422745) should contact the administrators of that study.
Supporting Information: Study Protocol, ICF
Time Frame: After completion of study
Access Criteria: Cosmos-Web Project Proposal Form Approved by Dr. Brickman

REFERENCES:
- [Background] Brickman AM, Khan UA, Provenzano FA, Yeung LK, Suzuki W, Schroeter H, Wall M, Sloan RP, Small SA. Enhancing dentate gyrus function with dietary flavanols improves cognition in older adults. Nat Neurosci. 2014 Dec;17(12):1798-803. doi: 10.1038/nn.3850. Epub 2014 Oct 26. PMID 25344629
- [Background] Hale C, Last BS, Meier IB, Yeung LK, Budge M, Sloan RP, Small SA, Brickman AM. The ModRey: An Episodic Memory Test for Nonclinical and Preclinical Populations. Assessment. 2019 Sep;26(6):1154-1161. doi: 10.1177/1073191117723113. Epub 2017 Aug 11. PMID 28799411
- [Background] Sloan RP, Wall M, Yeung LK, Feng T, Feng X, Provenzano F, Schroeter H, Lauriola V, Brickman AM, Small SA. Insights into the role of diet and dietary flavanols in cognitive aging: results of a randomized controlled trial. Sci Rep. 2021 Feb 15;11(1):3837. doi: 10.1038/s41598-021-83370-2. PMID 33589674
- [Derived] Vyas CM, Manson JE, Sesso HD, Cook NR, Rist PM, Weinberg A, Moorthy MV, Baker LD, Espeland MA, Yeung LK, Brickman AM, Okereke OI. Effect of multivitamin-mineral supplementation versus placebo on cognitive function: results from the clinic subcohort of the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial and meta-analysis of 3 cognitive studies within COSMOS. Am J Clin Nutr. 2024 Mar;119(3):692-701. doi: 10.1016/j.ajcnut.2023.12.011. Epub 2024 Jan 18. PMID 38244989
- [Derived] Yeung LK, Alschuler DM, Wall M, Luttmann-Gibson H, Copeland T, Hale C, Sloan RP, Sesso HD, Manson JE, Brickman AM. Multivitamin Supplementation Improves Memory in Older Adults: A Randomized Clinical Trial. Am J Clin Nutr. 2023 Jul;118(1):273-282. doi: 10.1016/j.ajcnut.2023.05.011. Epub 2023 May 24. PMID 37244291